CLINICAL TRIAL: NCT06269484
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Safety of Zibotentan/Dapagliflozin in Combination Compared to Zibotentan Monotherapy, Zibotentan/Dapagliflozin and Zibotentan Monotherapy Compared to Placebo in Participants With Cirrhosis
Brief Title: A Phase IIb Study to Evaluate the Safety of Zibotentan/Dapagliflozin in Participants With Cirrhosis-ZEAL-UNLOCK
Acronym: ZEAL UNLOCK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D4326C00004; 2023-506893-11-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2024-02-02; First posted 2024-02-21 (Actual); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Liver Cirrhosis
Keywords: Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — ZD4054; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Group 1 (Placebo Comparator): Participants will receive once daily dose of placebo matching zibotentan capsule + placebo matching dapagliflozin tablet for 6 weeks
  Interventions: Drug: Placebo (placebo matching zibotentan capsule and placebo matching dapagliflozin tablet)
- Treatment Group 2 (Experimental): Participants will receive once daily zibotentan capsule + placebo matching dapagliflozin tablet for 6 weeks
  Interventions: Drug: Zibotentan + placebo (placebo matching dapagliflozin tablet)
- Treatment Group 3 (Experimental): Participants will receive once daily zibotentan capsule + dapagliflozin tablet 10 mg for 6 weeks
  Interventions: Drug: Zibotentan + dapagliflozin

INTERVENTIONS:
Drug: Placebo (placebo matching zibotentan capsule and placebo matching dapagliflozin tablet) — placebo capsule (matching zibotentan capsule)
  placebo tablet (matching dapagliflozin tablet)
  Arms: Treatment Group 1
Drug: Zibotentan + placebo (placebo matching dapagliflozin tablet) — zibotentan capsule
  placebo tablet (matching dapagliflozin tablet)
  Arms: Treatment Group 2
Drug: Zibotentan + dapagliflozin — zibotentan capsule
  dapagliflozin 10 mg tablet
  Arms: Treatment Group 3

SUMMARY:
This is a Phase IIb multicentre, randomised, double-blind, parallel-group, placebo-controlled study to evaluate the safety of zibotentan/dapagliflozin in combination as compared to zibotentan monotherapy as well as zibotentan/dapagliflozin and zibotentan monotherapy as compared to placebo in patients with cirrhosis.

DETAILED DESCRIPTION:
The study is designed to evaluate the safety of zibotentan/dapagliflozin in combination as compared to zibotentan monotherapy as well as zibotentan/dapagliflozin in combination and zibotentan monotherapy as compared to placebo in patients with cirrhosis with or without a history of decompensation. The study will be conducted in approximately 52 study centers in North America, Asia and Europe.

ELIGIBILITY:
Inclusion Criteria:

≥ 18 and ≤ 80 years of age at the time of signing the informed consent.

Clinical and/or histological diagnosis of cirrhosis.

Note: Either history of decompensation or compensated cirrhosis with signs of CSPH, including varices at endoscopy or collaterals at imaging (within 12 months prior to screening), and/or liver stiffness using vibration controlled elastography, liver stiffness > 25 kPa or > 21 kPa, and platelets < 150 × 10^99 (at time of screening).

Model for end stage liver disease score (MELD) < 15.

Child-Pugh score < 10.

No ascites or ascites up to grade 2 without change in diuretic treatment within the last month prior to first dose of study intervention and no paracentesis within the last month.

No evidence of worsening of hepatic function (eg, no clinically significant change in signs, symptoms, or laboratory parameters of hepatic disease status) within the last month prior to dosing, as determined by the investigator or usual practitioner.

No current or prior (within 1 month of enrolment) medical treatment with an SGLT2 inhibitor or endothelin receptor antagonist.

On no or a stable dose of beta blockers, with no major dose changes within 1 month prior to the first dose of study intervention.

Males or females of non-childbearing potential:

Male participants must be surgically sterile, abstinent, or must use in conjunction with their female partner a highly effective method of contraception from the time they sign the informed consent document and for 3 months after the last dose of study intervention to prevent pregnancy in a partner. In addition, the male participant should use a condom for the duration of the study and for 3 months after the last dose of study intervention. Male participants must not donate or bank sperm during the same period.

Highly effective birth control methods are defined as those that can achieve a failure rate of less than 1% per year when used consistently and correctly.

Female participants must be of non-childbearing potential confirmed at screening by fulfilling one of the following criteria:

Post-menopausal: defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments; and also FSH levels in the post-menopausal range by central laboratory (Note: The post-menopausal range must be checked against the specific FSH assay used). In the absence of 12 months of amenorrhoea, a single FSH measurement is insufficient to define post-menopausal criteria. In case of perimenopause or infrequent periods with variable levels of FSH, women should be considered of childbearing potential and, therefore, not eligible for participation in this study.

Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.

Female participants must have a negative pregnancy test at screening and must not be lactating.

Capable of giving signed informed consent as described in Appendix A, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Provision of signed and dated, written ICF prior to any mandatory study-specific procedures, sampling, and analyses.

Provision of signed and dated written Optional Genomics Initiative Research Information and Consent Form prior to collection of samples for optional genomics initiative research that supports Genomic Initiative.

Exclusion criteria:

Any evidence of a clinically significant disease, which in the investigator's opinion makes it undesirable for the participant to participate in the study.

Alanine aminotransferase/transaminase or AST ≥ 150 U/L and/or total bilirubin

≥ 3 × ULN.

International normalised ratio > 1.7.

Serum/plasma levels of albumin ≤ 28 g/L.

Platelet count < 50 × 109L.

Acute kidney injury (AKI) within 3 months of screening.

History of encephalopathy of West Haven Grade 2 or higher

History of variceal haemorrhage within 6 months prior to screening.

Any history of hepatocellular carcinoma.

Any history of portal venous thrombosis.

Liver transplant or expected liver transplantation within 6 months of screening.

History of TIPS or a planned TIPS within 6 months from enrolment into the study.

Positive alcohol breath test or screen for drugs of abuse (excluding drugs prescribed by the participants' usual physician) at screening.

Ongoing or history of significant use of alcohol expected to preclude correct adherence to study procedures (For details, refer to Section 5.3.2).

Active treatment for HCV within the last 1 year or HBV anti-viral therapy for less than 1 year.

Active urinary tract infection or genital infection.

Uncontrolled diabetes mellitus (HbA1c > 8.5% or > 69 mmol/mol within the last month).

Participants with T1DM.

Renal transplant or chronic renal replacement therapy or short-term dialysis within the previous 6 months.

eGFR < 60 mL/min/1.73m2 (eGFRcr[AS]).

Acute coronary syndrome events within 3 months prior to screening.

Orthostatic hypotension or hypotension (systolic blood pressure < 95 mmHg or diastolic blood pressure < 60 mmHg).

New York Heart Association functional heart failure Class III or IV or patients with unstable heart failure requiring hospitalisation for optimisation of heart failure treatment and who are not yet stable on heart failure therapy within 6 months prior to screening.

Heart failure due to cardiomyopathies that would primarily require specific other treatment.

High output heart failure (eg, due to hyperthyroidism or Paget's disease).

Heart failure due to primary cardiac valvular disease/dysfunction, severe functional mitral or tricuspid valve insufficiency, or planned cardiac valve repair/replacement.

Participants treated with strong CYP3A4 inhibitor or strong or moderate CYP3A4 inducer within 14 days (St. John's Wort: 21 days) of study intervention administration; this includes grapefruit and grapefruit juice, if consumed more often than occasionally, or, in larger quantities.

History or ongoing allergy/hypersensitivity, as judged by the investigator, to SGLT2 inhibitors (eg, dapagliflozin, canagliflozin, empagliflozin), zibotentan, or drugs with a similar chemical structure to zibotentan.

Any clinically significant chronic disease or disorder (eg, cardiovascular, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, psychiatric, major physical impairment) which, as judged by the investigator, might put the participant at risk because of participation in the study, or probable alternative primary reason for participant's symptoms in judgment of investigator.

Acute liver injury caused by drug toxicity or by an infection.

Implanted electronic device such as pacemaker.

Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study centre).

Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

Male participant in a sexually active relation with pregnant or breastfeeding partner.

Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Exclusion Criteria for Participants Consenting to Optional Genetic Sampling:

Previous allogeneic bone marrow transplant.

Non-leukocyte depleted whole blood transfusion in 120 days of genetic sample collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (3):
  - Research Site, Englewood, Colorado
  - Research Site, Charleston, South Carolina
  - Research Site, San Antonio, Texas
- Australia (3):
  - Research Site, Adelaide
  - Research Site, Kogarah
  - Research Site, Mitcham
- Research Site, Mechelen, Belgium
- Czechia (3):
  - Research Site, Liberec
  - Research Site, Mladá Boleslav
  - Research Site, Prague
- Germany (2):
  - Research Site, Leipzig
  - Research Site, Tübingen
- Italy (3):
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
- Japan (7):
  - Research Site, Gifu
  - Research Site, Kawasaki-shi
  - Research Site, Kitakyusyu-shi
  - Research Site, Nagaoka-shi
  - Research Site, Niigata
  - Research Site, Sapporo
  - Research Site, Yokohama
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Mysłowice
  - Research Site, Poznan
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Nitra
  - Research Site, Trnava
- United Kingdom (5):
  - Research Site, Aberdeen
  - Research Site, Hull
  - Research Site, Ipswich
  - Research Site, London
  - Research Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: D4326C00004 Clinical Study Protocol v3.0 EU Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4326C00004&attachmentIdentifier=ca847da5-f0bc-41f0-b024-3a1ef456939f&fileName=D4326C00004_Clinical_Study_Protocol_v3.0_EU_Redacted.pdf&versionIdentifier=
- See also: D4326C00004 CSR Synopsis - Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4326C00004&attachmentIdentifier=e9591c1f-141b-4208-8506-ac74d2903b9e&fileName=D4326C00004_CSR_Synopsis_-_Redacted.pdf&versionIdentifier=
- See also: D4326C00004 Statistical Analysis Plan v2.0 Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4326C00004&attachmentIdentifier=5f1c273b-59d5-4802-ae09-25e87276675f&fileName=D4326C00004_Statistical_Analysis_Plan_v2.0_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on February 2024 and the last participant was enrolled in September 2024.
Pre-assignment Details: Of 88 study participants, 73 met inclusion criteria and were not withdrawn by subject and subsequently randomised to treatment.
Groups:
- Zibo/Dapa: Zibotentan capsule + dapagliflozin 10 mg
- Zibo: Zibotentan capsule + placebo
- Placebo: Placebo + placebo
Period: Overall Study
Arm/Group | Zibo/Dapa | Zibo | Placebo
Started (Number randomised) | 24 | 25 | 24
TREATED (Number started treatment) | 24 | 24 | 24
Completed | 20 | 24 | 22
Not Completed | 4 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 2
Not completed — All other reasons apart from specified | 1 | 0 | 0
Not completed — Randomised but not started treatment | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomised subjects who received at least one dose of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zibo/Dapa | Zibo | Placebo | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.2 (11.4) | 59.5 (8.9) | 62.6 (8.4) | 60.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 7 | 21
  Male | 18 | 16 | 17 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 1 | 8
  Not Hispanic or Latino | 20 | 21 | 23 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 4 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 20 | 20 | 20 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Subjects With Any of the Components of the Composite Endpoint: >2kg Increase in Body Weight (Office-based), >2 L Increase in Total Body Water, Increase in 2 or More Loop-diuretic Equivalents, Fluid Retention Adverse Event (AE)
Description: Cumulative number of subjects with event of composite fluid retention endpoint
Time Frame: baseline to Week 6
Population: All randomised subjects who received at least one dose of treatment are included in the analysis.
  For intercurrent events treatment policy strategy was used. No imputation was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 24 | 24 | 24
Participants | 14 | 14 | 6
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Proportions used for comparison; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Risk Difference (RD) = 0, 90% CI 2-sided [-0.24 to 0.24] — Risk difference for proportions presented. The associated CI is the exact unconditional 90% (two-sided) computed based on score statistic
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Proportions used for comparison; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Risk Difference (RD) = 0.33, 90% CI 2-sided [0.09 to 0.55] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Proportions used for comparison; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Risk Difference (RD) = 0.33, 90% CI 2-sided [0.09 to 0.55] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Body Weight
Description: Change in site body weight
Time Frame: at Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 20 | 24 | 22
kg | -1.08 [-1.88 to -0.28] | 0.64 [-0.11 to 1.39] | -0.53 [-1.31 to 0.24]
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -1.72, 90% CI 2-sided [-2.82 to -0.62]
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -0.55, 90% CI 2-sided [-1.66 to 0.56]
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 1.17, 90% CI 2-sided [0.09 to 2.25]

3. Secondary Outcome: Change From Baseline in Body Fat Mass
Time Frame: at Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 20 | 24 | 22
kg | -1.68 [-2.43 to -0.94] | -0.23 [-0.93 to 0.48] | -0.30 [-1.03 to 0.42]
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -1.45, 90% CI 2-sided [-2.48 to -0.43]
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -1.38, 90% CI 2-sided [-2.42 to -0.34]
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 0.07, 90% CI 2-sided [-0.94 to 1.09]

4. Secondary Outcome: Change From Baseline in Total Body Water
Time Frame: at Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 20 | 24 | 22
L | 0.36 [-0.22 to 0.94] | 0.66 [0.12 to 1.21] | -0.36 [-0.92 to 0.21]
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -0.30, 90% CI 2-sided [-1.10 to 0.49]
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 0.72, 90% CI 2-sided [-0.09 to 1.52]
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 1.02, 90% CI 2-sided [0.23 to 1.81]

5. Secondary Outcome: Change From Baseline in Extracellular Water Volume
Time Frame: at Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 20 | 24 | 22
L | 0.38 [0.09 to 0.66] | 0.38 [0.11 to 0.65] | -0.15 [-0.43 to 0.13]
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 0, 90% CI 2-sided [-0.40 to 0.39]
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 0.53, 90% CI 2-sided [0.12 to 0.93]
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 0.53, 90% CI 2-sided [0.14 to 0.92]

6. Secondary Outcome: Change From Baseline in Intracellular Water Volume
Time Frame: at Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: L
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 20 | 24 | 22
L | 0.08 [-0.24 to 0.40] | 0.30 [0 to 0.60] | -0.19 [-0.50 to 0.12]
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -0.22, 90% CI 2-sided [-0.66 to 0.22]
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 0.27, 90% CI 2-sided [-0.18 to 0.71]
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 0.49, 90% CI 2-sided [0.05 to 0.92]

7. Secondary Outcome: Change in Body Weight (kg) Over Time Course of Study
Description: Change in home body weight
Time Frame: at Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 16 | 20 | 15
kg | -1.754 [-2.541 to -0.967] | 0.021 [-0.692 to 0.734] | -1.256 [-2.077 to -0.435]
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -1.775, 90% CI 2-sided [-2.836 to -0.714]
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -0.499, 90% CI 2-sided [-1.637 to 0.639]
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 1.277, 90% CI 2-sided [0.183 to 2.371]

8. Secondary Outcome: Change in Total Dosage of Loop-diuretic Equivalents Use
Description: One loop-diuretic equivalent = 40 mg furosemide = 1 mg bumetanide = 20 mg torsemide = 50 mg ethacrynic acid. In Japan, one loop-diuretic equivalent = 40 mg furosemide = 8 mg torsemide = 60 mg azosemide.
Time Frame: at Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Loop-diuretic *mg* equivalent
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 20 | 24 | 22
Loop-diuretic *mg* equivalent | 1.282 [-2.045 to 4.609] | 6.340 [3.104 to 9.576] | 1.338 [-1.953 to 4.629]
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -5.058, 90% CI 2-sided [-9.700 to -0.417] — Note: Model assumption was violated due to skewed data distribution and the results should not be interpreted
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -0.056, 90% CI 2-sided [-4.736 to 4.624] — Note: Model assumption was violated due to skewed data distribution and the results should not be interpreted
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = 5.002, 90% CI 2-sided [0.388 to 9.617] — Note: Model assumption was violated due to skewed data distribution and the results should not be interpreted

9. Secondary Outcome: Cumulative Number of Subjects With Either of the Two Components of This Composite: 1. >3 L Increase in Total Body Water Volume From Baseline to Week 6 2. Increase in 3 or More Loop-diuretics Equivalents Use
Description: Cumulative number of subjects with event of composite and the components of total body water and total dosage of loop-diuretic equivalents
Time Frame: from baseline to Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 24 | 24 | 24
Participants | 7 | 9 | 2
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Proportions used for comparison; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Risk Difference (RD) = -0.08, 90% CI 2-sided [-0.31 to 0.15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Proportions used for comparison; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Risk Difference (RD) = 0.21, 90% CI 2-sided [0.02 to 0.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Proportions used for comparison; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Risk Difference (RD) = 0.29, 90% CI 2-sided [0.09 to 0.49] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Absolute Change in Systolic Blood Pressure
Time Frame: at Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mmHg
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 21 | 24 | 22
mmHg | -12.0 [-16.1 to -7.9] | -2.6 [-6.5 to 1.2] | -0.1 [-4.1 to 3.9]
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -9.4, 90% CI 2-sided [-15.0 to -3.8]
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -11.9, 90% CI 2-sided [-17.7 to -6.1]
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -2.5, 90% CI 2-sided [-8.1 to 3.0]

11. Secondary Outcome: Absolute Change in Diastolic Blood Pressure
Time Frame: at Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mmHg
Arm/Group | Zibo/Dapa | Zibo | Placebo
Number analyzed (Participants) | 21 | 24 | 22
mmHg | -9.1 [-11.3 to -6.8] | -2.5 [-4.7 to -0.3] | 1.8 [-0.5 to 4.0]
Statistical Analysis 1: Comparison: Zibo/Dapa vs Zibo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -6.5, 90% CI 2-sided [-9.7 to -3.4]
Statistical Analysis 2: Comparison: Zibo/Dapa vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -10.8, 90% CI 2-sided [-14.1 to -7.6]
Statistical Analysis 3: Comparison: Zibo vs Placebo; Test type: Other — No test was performed; Mixed Models Analysis; Comparisons are done as Zibo adjusted Zibo/Dapa, Placebo adjusted Zibo/Dapa or Placebo adjusted Zibo; Mean Difference (Net) = -4.3, 90% CI 2-sided [-7.4 to -1.1]

ADVERSE EVENTS:
Time Frame: Adverse events reported are adverse events with an onset date on or after the date of first dose of IP and until end of study for each participant which in general was 6 weeks treatment period and 2 weeks follow-up period.
Arm/Group | Zibo/Dapa | Zibo | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24 | 2/24 | 1/24
Other Adverse Events (participants affected / at risk) | 14/24 | 15/24 | 4/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zibo/Dapa (N=24) | Zibo (N=24) | Placebo (N=24)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zibo/Dapa (N=24) | Zibo (N=24) | Placebo (N=24)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 6 (7) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 3 (5) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 5 (7) | 1 (1)
Weight increased (Investigations) | 2 (3) | 3 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding study results for a period that is less than or equal to 60 days from the date that the communication is submitted to the sponsor for review. The sponsor can require changes to the communication but cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT06269484/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT06269484/SAP_001.pdf